CLINICAL TRIAL: NCT01019993
Title: Prospective Study of the Effects of Non-dependent Lung High Frequency Positive Pressure Ventilation on the Right Ventricular Function for Thoracotomy
Brief Title: Non-dependent Lung High Frequency Positive Pressure Ventilation (HFPPV) and Right Ventricular Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Mohamed R. El-Tahan, M.D, Anaesthesia and Surgical ICU, Faculty of Medicine, Mansoura University, Egypt (current affiliation: Department of Anaesthesia and Surgical ICU, Faculty of Medicine, King Faisal University, Dammam, KSA)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39-01-2004
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Lung Diseases; Esophageal Diseases
Keywords: Thoracotomy; one lung ventilation; HFPPV; right ventricular function.
MeSH Terms: conditions — Lung Diseases; Esophageal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- good pulmonary functions (group N) (Active Comparator): The patients were allocated if they have forced vital capacity (FVC %) and/or forced expiratory volume in 1 sec (FEV1%) of 80% of predicted or more
  Interventions: Procedure: conventional OLV followed with IL-HFPPV
- pulmonary dysfunction (group PD) (Active Comparator): The patients were allocated if they have FVC and/or FEV1 of 50%-79% of predicted
  Interventions: Procedure: conventional OLV followed with IL-HFPPV

INTERVENTIONS:
Procedure: conventional OLV followed with IL-HFPPV — The patients' lungs were mechanically ventilated with intermittent positive pressure ventilation using fraction of inspired oxygen (FiO2) of 0.5 in air, tidal volume (VT) of 8 mL/kg, inspiratory to expiratory [I: E] ratio of 1:2.5, zero positive end-expiratory pressure (PEEP), respiratory rate (R.R) was adjusted to achieve an arterial carbon dioxide tension (PaCO2) 35-45 mm Hg and peak inspiratory pressures were limited to 35 cm H2O. After pleurotomy, OLV was initiated with the same ventilatory settings for the dependent lung. After 30 min, the non-dependent collapsed lung was ventilated using HFPPV mode (IL-HFPPV) with another identical ventilator, with an internal circuit of low compliance, using FiO2 of 0.5 in air, VT 3 mL/kg, I: E ratio <0.3 and R.R 60 breaths/min.
  Other Names: KONTRON ABT 5300 ventilator, UK

SUMMARY:
The investigators hypothesized that the application of volume-controlled HFPPV to the non-dependent lung during one-lung ventilation (OLV) for thoracotomy in patients with good pulmonary functions and mild-to-moderate pulmonary dysfunction may provide preservation of the right ventricular (RV) function, adequate oxygenation and optimum surgical conditions.

The investigators evaluated the effects of IL-HFPPV on RV ejection fraction (REF), RV end-diastolic volume (RVEDVI), RV stroke work (RVSWI), pulmonary vascular resistance (PVRI), and stroke volume (SVI) indices, oxygen delivery (DO2) and uptake (VO2), shunt fraction (Qs: Qt), and surgical field conditions during OLV for thoracotomy in patients with good and mild-to-moderate impaired pulmonary functions.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) provides an adequate operative field, but is opposed by the induced hypoxic pulmonary vasoconstriction (HPV) in the non-ventilated lung. It may preserve overall oxygen delivery, however with deleterious increase in shunt fraction and pulmonary vascular resistance.1-2Right ventricular (RV) overload resulting from these increases in its afterload influences postoperative morbidity and mortality. Intrinsic positive end-expiratory pressure (PEEPi) occurs frequently during OLV for thoracic surgery in the dependent lung of patients with pulmonary hyperinflation as opposed to patients with normal pulmonary function.3 The different approaches for the correction of hypoxemia during OLV may require some degree of recruitment of the non-dependent lung (IL), with different maneuvers such as the application of continuous positive pressure ventilation (CPAP) or high frequency jet ventilation (HFJV) to the non-dependent lung. These recruitment strategies, although they may improve arterial saturation, may concurrently decrease cardiac output, therefore having contradictory effects on overall oxygen delivery.4-6 Gas trapping may occur with increased ventilatory frequency during HFJV. This may impair RVEF through the increases in RV afterload.7 Therefore, the use of high frequency positive pressure ventilation (HFPPV) using tidal volumes just greater than the dead space increases arterial oxygen tension (PaO2) and the carbon dioxide excretion (VCO2) linearly with increasing peak airway pressure.8 We hypothesized that the application of volume-controlled HFPPV to the non-dependent lung during OLV for thoracotomy in patients with good pulmonary functions and mild-to-moderate pulmonary dysfunction may provide preservation of the RV function, adequate oxygenation and optimum surgical conditions.

We evaluated the effects of IL-HFPPV on RV ejection fraction (REF), RV end-diastolic volume (RVEDVI), RV stroke work (RVSWI), pulmonary vascular resistance (PVRI), and stroke volume (SVI) indices, oxygen delivery (DO2) and uptake (VO2), shunt fraction (Qs: Qt), and surgical field conditions during OLV for thoracotomy in patients with good and mild-to-moderate impaired pulmonary functions.

ELIGIBILITY:
Inclusion Criteria:

* Thirty-three patients ASA physical status II-III) scheduled for elective open thoracic surgery were prospectively included in this study at the authors' cardiothoracic center. Approval of the institutional ethical committee and informed written consent was obtained specifically for use of pulmonary artery catheter which is not routinely used in thoracic procedures at the authors' center.

Exclusion Criteria:

* Patients with decompensated cardiac (> New York Heart Association II), pulmonary (vital capacity or FEV1% < 50% of the predicted values), hepatic, and renal diseases, arrhythmias, pulmonary hypertension (mean pulmonary artery pressure (MPAP) > 30 mm Hg), and previous history of pneumonectomy, bilobectomy or lobectomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome variables included right ventricular function (REF, RVEDVI, and RVSWI). | before (Baseline) and10 min after induction of anesthesia during two-lung ventilation, 15 and 30 min after OLV, 15, 30, 60 min after IL-HFPPV, and 15 min after resuming of two-lung ventilation (TLV

SECONDARY OUTCOMES:
Secondary outcome variables were hemodynamic parameters (HR, MAP, CI, SVI, and PVRI), oxygenation parameters (DO2, VO2, and Qs:Qt) and surgical field conditions. | before (Baseline) and10 min after induction of anesthesia during two-lung ventilation, 15 and 30 min after OLV, 15, 30, 60 min after IL-HFPPV, and 15 min after resuming of two-lung ventilation (TLV)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D., Principal Investigator — Anaesthesia and Surgical ICU, Faculty of Medicine, Mansoura University, Egypt (current affiliation: Department of Anaesthesia and Surgical ICU, Faculty of Medicine, King Faisal University, Dammam, KSA; Reda A. Hamad, M.D., Study Chair — Cardiothoracic Unit, Faculty of Medicine, Mansoura University, Egypt (current affiliation: Prince Sultan Cardiac Centre, Riyadh, KSA
Locations (1):
- Cardiothoracic Unit, Faculty of Medicine, Mansoura University, Egypt, Al Mansurah, DK, Egypt